CLINICAL TRIAL: NCT04778085
Title: Young People's Experiences of Illness Management and Recovery (IMR) - an Explorative Study
Brief Title: Young People and Illness Management and Recovery (IMR)
Status: Terminated | Type: Observational
Why Stopped: As anticipated by the protocol
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Anne-Lise Holmesland, Prinsipal investigator, University Hospital, Akershus
Other Study IDs: 20/09657
Record Dates: First submitted 2021-02-14; First posted 2021-03-02 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Psychosis; Bipolar Disorder; Other Diagnoses and Conditions
Keywords: Psychosis
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder | interventions — Salvage Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMR patients: Patients from outpatient clinics receiving IMR from trained IMR therapists and IMR therapists in training.
  Interventions: Behavioral: Illness management and recovery
- IMR therapists and other staff: Clinic leaders, IMR therapists and other staff participating in semi-structured individual or group interviews.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Behavioral: Illness management and recovery — Treatment given in groups, weekly for 10-12 months.
  Other Names: IMR
  Groups: IMR patients
Other: Semi-structured interviews — Semi-structured individual or group interviews conducted three times with staff on each participating outpatient clinic.
  Groups: IMR therapists and other staff

SUMMARY:
The study is a combined clinical patient outcome study and a health-services research sub-study. Illness management and recovery (IMR) constitutes an evidence-based practice with 11 modules focusing on personal recovery developed for adults with severe mental health illnesses. IMR can be offered in groups or individually, once a week for 10-12 months.

Little is known about how young people experience the utility of IMR treatment groups in child and adolescent mental health outpatient clinics. The primary aim is to explore in-depth how the participants experience the utility of the IMR approach. The health research sub-study will provide new insights into the IMR implementation process in outpatient clinics for adolescents.

DETAILED DESCRIPTION:
IMR has previously been implemented for adolescents in an inpatient unit in the hospital's catchment area. In order to offer the same treatment to all young patients, IMR treatment groups will be established in 4 out of 7 outpatient clinics in the hospital's catchment area. Participants belonging to the clinics in which no IMR treatment groups are being established will be invited to participate in IMR groups in clinics nearby.

The primary aim is to gain new insight into how young people experience the utility of IMR treatment groups conducted in outpatient practices and, if relevant, which changes could be made to adapt IMR more to young people. To explore how the participants experience the utility of IMR treatment groups, a qualitative focus-group study, consisting of a maximum of 5 focus-group interviews will be conducted. The participants in each IMR treatment group will be offered treatment once a week up to 10-12 months. To establish an IMR treatment group a minimum of 4 patients and a maximum of 8 participants must participate. Participants are mainly being included in the IMR treatment groups at the two primary admissions to each treatment group. Thus, some of the participants in the focus-groups may have participated in IMR groups for less than 10-12 months.

Secondary outcomes are related to fidelity to the model and the extent to which IMR treatment groups are implemented at an organizational level. The treatment groups will be led by trained IMR-therapists employed in inpatient units, together with therapists in training who are employed in outpatient clinics. Leaders and other clinicians in the outpatient clinics will contribute knowledge about the extent to which core components of IMR are being implemented, as well as information relating to quality improvement and individual adjustment. Two of the out-patient clinics in which no IMR group is being established will be included in the sub-study. The clinics will receive written feedback after each measurement time to support quality improvement.

The goal is to include up to 48 participants receiving IMR treatment in outpatient clinics. Up to 8 hospitalized participants will participate in a pilot focus-group interview. In the sub-study, a maximum of 16 IMR therapists, trained and in training, and up to 24 staff members will be invited to participate.

ELIGIBILITY:
Inclusion Criteria Patients:

Outpatient units:

* Included in the IMR group in one of the outpatient clinics
* Able to give informed consent

Inpatient unit (focus group):

* 13-17 years of age
* Current or previous patient
* Able to understand and speak Norwegian
* Able to give informed consent

Exclusion criteria (inpatient unit)

* Younger than 13 years
* Mental retardation
* Manic phase

Inclusion Criteria: IMR therapists:

* IMR therapist leading IMR treatment groups in one of the participating outpatient clinics
* Trained or training in IMR
* Employed at the Department for Child and Adolescent Mental Health Services at Akershus University Hospital.

Inclusion Criteria: Other staff members

• Employed at the Department for Child and Adolescent Mental Health Services at Akershus University Hospital.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients between 13-17 years of age suffering from or having symptoms of psychosis or bipolar disorders, and who participate in an IMR treatment group at one of the 4 (out of 7) outpatient clinics in the hospitals catchment area, and who are able to give informed consent. Up to 8 inpatients or previous inpatients between 13- 17 years of age suffering from various diagnoses will be invited to participate in a pilot focus-group interview. Trained clinicians and clinicians in training contribute to the implementation in the outpatient clinics together with clinic leaders and other clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Focus-group interview aiming to explore the significance of the participant's own understanding of and knowledge about the disorder. | End of treatment group, on average 11 months.
  Focus-group interviews when the treatment group has come to an end aimed at exploring different perspectives on IMR treatment.
Focus-group interview aiming to explore the impact of the IMR treatment on dealing with everyday life. | End of treatment group, on average 11 months.
  Focus-group interviews when the treatment group has come to an end aimed at exploring different perspectives on IMR treatment.
Focus-group interview aiming to explore the importance of meeting other young people in the same situation. | End of treatment group, on average 11 months.
  Focus-group interviews when the treatment group has come to an end aimed at exploring different perspectives on IMR treatment.

SECONDARY OUTCOMES:
The Illness Management and Recovery Scale (IMRS) | Baseline (0 months), 6 and 12 months.
  A 15-item scale that assesses illness self-management on a 5-point Likert scale where 5 indicates full self-management and 0 indicates no self-management. The scale measures consumer behavior relating to core components in the IMR program. The scale includes parallel clinician and consumer versions. Participants participating in IMR groups for less than 10-12 months will attend fewer measuring times.
The Illness Management Fidelity Scale | Baseline (0 months), 6 and 12 months.
  Assesses the degree of fidelity with 13 items on a 5-point Likert scale where 5 indicates full implementation and 0 indicates no implementation. Filled in by researchers on the basis of a semistructured interview with staff members.
General Organizational Index | Baseline (0 months), 6 and 12 months.
  A 12-item scale measuring organizational outcome of implementation, on a 5-point Likert scale where 5 indicates full implementation and 0 indicates no implementation. The scale is filled in by researchers on the basis of a semi-structured interview with staff members.
Attendance registration | Baseline (0 months), 3, 6, 9 and 12 months.
  The number of sessions the patients are attending in the IMR treatment group.

OTHER OUTCOMES:
Mapping the total number of patients identified receiving a psychosis-related diagnosis within the categories F 20-39 (ICD 10) for the years 2021-2023. | End of treatment group, on average of 11 months.
  The numbers will be displayed in the form of statistics obtained in the hospital. The numbers will be compared to what has been reported in the annual reports for the clinics from 2015 to 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Holmesland, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus universitetssykehus, Viken, Norway

IPD SHARING:
Plan to Share IPD: No